CLINICAL TRIAL: NCT05888454
Title: Dando Pasos Juntos: An Integrative Group Program for Type 2 Diabetes Mellitus
Brief Title: Integrative Group Program for Type 2 Diabetes Mellitus (T2DM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TecSalud Investigación Clínica (Other)
Collaborators: TecSalud (Unknown); Fundación Santos y de la Garza Evia I.B.P (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dando pasos juntos
Record Dates: First submitted 2023-05-15; First posted 2023-06-05 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Integrative Medicine; Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Conventional treatment for T2DM + Integrative Group Program
  Interventions: Other: Integrative Group Program; Other: Conventional treatment for T2DM
- Control Group (Active Comparator): Conventional treatment for T2DM
  Interventions: Other: Conventional treatment for T2DM

INTERVENTIONS:
Other: Integrative Group Program — The integrative group program consists of 6 in-person sessions directed by a health coach and occurring every other week, and 6 asynchronous educative sessions during a period of 12 weeks.
  Arms: Experimental Group
Other: Conventional treatment for T2DM — Conventional medical treatment for T2DM

SUMMARY:
This is an open, randomized, controlled trial to determine the impact of an integrative group program on metabolic control and wellbeing perception of patients with T2DM. The integrative group program consists of 6 in-person sessions directed by a health coach and occurring every other week, and 6 asynchronous educative sessions during a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* T2DM diagnosis of less than 5 years
* Age 18 to 80 years
* Current residence in Nuevo León, México
* Availability to attend in-person sessions
* Provides written informed consent
* Able to read and write

Exclusion Criteria:

* Currently under insulin treatment
* T2DM diagnosis more than 5 years ago
* Comorbidities such as active cancer, acquired immunodeficiency (HIV+, AIDS), liver, cardiovascular, renal, pulmonary or thyroid disease.
* History of severe neurologic or psychiatric disease (current or past diagnosis)
* Currently pregnant or intention of pregnancy in the following 3 months
* Males that consume more than 4 alcoholic beverages daily or 14 weekly
* Females that consume more than 3 alcoholic beverages daily or 7 weekly
* Consumption of any illicit drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
HbA1c levels (%) | Baseline to 12 weeks

SECONDARY OUTCOMES:
HbA1c levels (%) | Baseline to 12 weeks and 36 weeks
Fasting insulin (mU/mL) | Baseline to 12 weeks and 36 weeks
Fasting glucose (mg/dL) | Baseline to 12 weeks and 36 weeks
Homeostatic Model Assessment (HOMA index) | Baseline to 12 weeks and 36 weeks
High-sensitivity C-reactive protein (hs-CRP, mg/dL) | Baseline to 12 weeks and 36 weeks
Change in lifestyle instrument | Baseline to 12 weeks and 36 weeks
  Instrument to measure diabetic lifestyles (IMEVID) total score
Subjective sense of wellbeing instrument | Baseline to 12 weeks and 36 weeks
  Positive emotion, Engagement, Relationships, Meaning, and Accomplishment (PERMA-profiler) score
Adherence to pharmacological interventions for T2DM | Baseline to 12 weeks and 36 weeks
  Adherence to Refill and Medication Scale (ARMS) score
Change in dose of pharmacological interventions for T2DM | Baseline to 12 weeks and 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tania Zertuche, MD, Principal Investigator — Director de Instituto de Bienestar y Prevención
Locations (2):
- Mexico (2):
  - Centro Médico Zambrano Hellion, Fundación Santos y de la Garza Evia I.B.P, TecSalud, San Pedro Garza García, Nuevo León
  - Centro de Salud Integral, Fundación Santos y de la Garza Evia I.B.P, TecSalud, Santa Catarina, Nuevo León

IPD SHARING:
Plan to Share IPD: No